CLINICAL TRIAL: NCT04235036
Title: Phase II Trial Evaluating the Safety and Efficacy of Combined CD20- and BTK-Targeted B Cell Depleting Therapy With Rituximab and Ibrutinib in the Primary Treatment of Chronic Graft-Versus-Host Disease
Brief Title: Ibrutinib and Rituxan for Chronic GVHD
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Low Recruitment
Sponsor: Northside Hospital, Inc. (Other)
Collaborators: Pharmacyclics LLC. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NSH 1219
Record Dates: First submitted 2019-08-19; First posted 2020-01-21 (Actual); Results first posted 2024-12-13 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-12

CONDITIONS: Graft Vs Host Disease
Keywords: ibrutinib; rituximab; cGVHD; chronic GVHD
MeSH Terms: conditions — Graft vs Host Disease; Bronchiolitis Obliterans Syndrome | interventions — Rituximab; ibrutinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Rituximab + Ibrutinib (Experimental): Eligible patients will be those with a first episode of symptomatic cGVHD, requiring systemic immunosuppression for control of symptoms. Following study entry, patients will be started on rituximab plus ibrutinib.
  Interventions: Drug: Rituximab; Drug: Ibrutinib

INTERVENTIONS:
Drug: Rituximab — Rituximab is given IV weekly x 4 weeks (to be started on study day 7 ± 3 days), then IV q3months x 4 doses (months 4, 7, 10, 13).
Drug: Ibrutinib — Ibrutinib is given orally every day (28-day cycles) for a total of 12 cycles.

SUMMARY:
This is a phase II trial evaluating the safety and efficacy of the combination of Ibrutinib and Rituximab as primary treatment of chronic GVHD. We plan to enroll 35 patients on this study. Patients will be formally monitored monthly for 12 months to evaluate for outcome and safety endpoints. All other assessments will be done at the physician's discretion or institutional standards. All patients, responders and treatment failures, will be followed for a period of one year from the time of initiation of therapy. The primary endpoint will be the proportion of patients that are alive and off all systemic IST at 12 months following initiation of treatment.

ELIGIBILITY:
Inclusion Criteria:

* First episode of systemic immunosuppression-requiring cGVHD, defined as classic or overlap cGVHD by the NIH consensus criteria.
* Previously untreated cGVHD, defined by having received <10 days of corticosteroids or alternative systemic immunosuppressive agent started specifically for a new diagnosis of cGVHD.
* KPS 70% or greater

Exclusion Criteria:

* Late persistent or recurrent acute GVHD
* Active uncontrolled infection
* History of HIV infection; active HBV or HCV infection
* Inability to tolerate oral medications
* Progressive or recurrent malignancy following allogeneic transplant
* Exposure to BTK inhibitor following transplant
* Received prior treatment with ECP for cGVHD

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2019-12-16 (Actual); Primary Completion 2022-12-23 (Actual); Study Completion 2022-12-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scott R Solomon, MD, Principal Investigator — Northside Hospital
Locations (1):
- Northside Hospital, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Rituximab + Ibrutinib
Started | 15
Completed | 15
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Rituximab + Ibrutinib
Number analyzed (Participants) | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 11
  >=65 years | 4
Age, Continuous [Median (Full Range); unit: years] | 58 [27 to 73]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 7
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 15

OUTCOME MEASURES:

1. Primary Outcome: The Number of Patients Who Remain Off Immunosuppressive Therapy at 12 Months After the Initiation of Treatment.
Description: The primary objective is to evaluate the efficacy of the combination of rituximab and ibrutinib versus the historical experience with rituximab alone in the upfront treatment of cGVHD. Patients will be followed for 12 months following the initiation of treatment to see if they remain off immunosuppressive therapy.
Time Frame: 12 months following initiation of treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Rituximab + Ibrutinib
Number analyzed (Participants) | 15
Participants | 4

2. Secondary Outcome: The Number of Patients Who Respond to Treatment Assessed by NIH Response Criteria Working Group Report.
Description: To estimate chronic GVHD response (CR + PR, both individual organ response and overall response, according to 2014 NIH Response Criteria Working Group Report [CR - resolution of all manifestations in each organ or site; PR - improvement in at least 1 organ or site without progression in any other organ or site])
Time Frame: 12 months following initiation of treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Rituximab + Ibrutinib
Number analyzed (Participants) | 15
Participants | 11

3. Secondary Outcome: How Long it Takes for Patients to Discontinue Treatment Defined as the Date All Systemic Immunosuppressive Therapy is Discontinued After Resolution of GVHD.
Description: To estimate time to discontinuation of systemic immunosuppression (defined as the date that all systemic IST has been discontinued after resolution of all reversible manifestations of cGVHD).
Time Frame: Up to 32 months
Measure: Median (Full Range); unit: months
Arm/Group | Rituximab + Ibrutinib
Number analyzed (Participants) | 15
months | 15 [0 to 31]

4. Secondary Outcome: How Many Patients Are Still Alive Without the Requirement for Second-line cGVHD Therapy Measured by Overall Survival at 12 Months Following the Initiation of Treatment.
Description: To estimate failure-free survival (defined as being alive without the requirement for second-line cGVHD therapy).
Time Frame: 12 months following initiation of treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Rituximab + Ibrutinib
Number analyzed (Participants) | 15
Participants | 7

5. Secondary Outcome: How Many Patients Have Not Relapsed Measured by Progression-free Survival at 12 Months Following the Initiation of Treatment.
Description: To estimate non-relapse mortality
Time Frame: 12 months following initiation of treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Rituximab + Ibrutinib
Number analyzed (Participants) | 15
Participants | 11

6. Secondary Outcome: How Many Patients Have Not Died Measured by Overall Survival at 12 Months Following the Initiation of Treatment.
Description: To estimate overall survival
Time Frame: 12 months following initiation of treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Rituximab + Ibrutinib
Number analyzed (Participants) | 15
Participants | 13

7. Secondary Outcome: Number of Patients With Treatment-related Adverse Events Grade 3 or Greater as Assessed by CTCAE v.4.0.
Description: To estimate the incidence of grade 3 or greater adverse events, possibly or probably related to either ibrutinib and/or rituximab.
Time Frame: 12 months following initiation of treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Rituximab + Ibrutinib
Number analyzed (Participants) | 15
Participants | 9

8. Secondary Outcome: Number of Patients With Treatment-related Adverse Events Total as Assessed by CTCAE v.4.0.
Description: To evaluate the safety and tolerability of combination of rituximab and ibrutinib versus the historical experience with rituximab alone in the upfront treatment of cGVHD.
Time Frame: 12 months following initiation of treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Rituximab + Ibrutinib
Number analyzed (Participants) | 15
Participants | 13

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | Rituximab + Ibrutinib
All-Cause Mortality (participants affected / at risk) | 2/15
Serious Adverse Events (participants affected / at risk) | 4/15
Other Adverse Events (participants affected / at risk) | 15/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rituximab + Ibrutinib (N=15)
Right hepatic hematoma (Blood and lymphatic system disorders) | 1 (1)
Right hepatic mass (Blood and lymphatic system disorders) | 1 (1)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
CMV colitis (Gastrointestinal disorders) | 1 (1)
Fever (Investigations) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rituximab + Ibrutinib (N=15)
COVID-19 Infection (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 2 (2)
Thrombocytopenia (Blood and lymphatic system disorders) | 7 (7)
Increased ALT (Metabolism and nutrition disorders) | 3 (3)
Lymphopenia (Blood and lymphatic system disorders) | 9 (9)
Leukopenia (Blood and lymphatic system disorders) | 9 (9)
Neutropenia (Blood and lymphatic system disorders) | 8 (8)
Increased AST (Metabolism and nutrition disorders) | 4 (4)
Hypertension (Cardiac disorders) | 3 (3)
Nose bleed (Blood and lymphatic system disorders) | 1 (1)
Hypocalcemia (Metabolism and nutrition disorders) | 4 (4)
Blurred vision (Eye disorders) | 1 (1)
Skin tightness (Skin and subcutaneous tissue disorders) | 1 (1)
Bacteremia (Infections and infestations) | 2 (2)
Mouth sores (Gastrointestinal disorders) | 3 (3)
Anemia (Blood and lymphatic system disorders) | 7 (7)
Hypergylcemia (Metabolism and nutrition disorders) | 6 (6)
Anorexia (Gastrointestinal disorders) | 2 (2)
Muscle pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Increased GGT (Metabolism and nutrition disorders) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 3 (3)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 3 (3)
Nausea (Gastrointestinal disorders) | 5 (5)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1)
Increased alkaline phosphatase (Metabolism and nutrition disorders) | 3 (3)
Myalgias (Musculoskeletal and connective tissue disorders) | 1 (1)
Right upper lip laceration (Skin and subcutaneous tissue disorders) | 1 (1)
Weight loss (Metabolism and nutrition disorders) | 2 (2)
Hypomagnesemia (Metabolism and nutrition disorders) | 3 (3)
Chest tightness (Cardiac disorders) | 1 (1)
Chills (Infections and infestations) | 2 (2)
Fever (Infections and infestations) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Hypotension (Cardiac disorders) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 4 (4)
Orthopnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 4 (4)
Taste alterations (Gastrointestinal disorders) | 1 (1)
Fatigue (General disorders) | 3 (3)
Headache (General disorders) | 1 (1)
Pericardial effusion (Cardiac disorders) | 1 (1)
Early satiety (Gastrointestinal disorders) | 2 (2)
Anal pain (Gastrointestinal disorders) | 1 (2)
Dry eyes (Eye disorders) | 1 (1)
Bruising (Blood and lymphatic system disorders) | 3 (3)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 2 (2)
Bilateral lower extremity edema (Cardiac disorders) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
C. diff infection (Infections and infestations) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Pharyngitis (Gastrointestinal disorders) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1)
Alopecia (General disorders) | 1 (1)
Urinary frequency (Renal and urinary disorders) | 1 (1)
Hypopigmentation (Skin and subcutaneous tissue disorders) | 1 (1)
Bilateral toe paronychia (Infections and infestations) | 1 (1)
Cellulitis (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-08-12): https://cdn.clinicaltrials.gov/large-docs/36/NCT04235036/Prot_SAP_000.pdf